CLINICAL TRIAL: NCT01778686
Title: Evaluation of [11C]Cimbi-36 as an Agonist PET Radioligand for Imaging of 5-HT2A Receptors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gitte Moos Knudsen (Other)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Professor, DMSc, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2012-002056-16
Record Dates: First submitted 2013-01-11; First posted 2013-01-29 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Positron Emission Tomography; Serotonin; 5-HT2A; Radioligand
MeSH Terms: interventions — Citalopram; Pindolol; Tryptophan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Citalopram and Pindolol (Experimental): Citalopram intravenous infusion starting 30 min before scanning, 40 mg/h for 1 hour.
  Pindolol peroral administration starting 3 days before scanning:
  Day 1: 2.5 mg 3 times daily, day 2: 5 mg 3 times daily, day 3: 7.5 mg 3 times daily, Day 4 (scan day) 7.5 mg morning and noon.
  Interventions: Drug: Citalopram and Pindolol
- Placebo (Placebo Comparator): Placebo for pindolol: sugar tablets that resembles pindolol
  Placebo for ATD: amino acid drink balanced formula (containing tryptophan)
  Placebo for Seropram: NaCl infusion
  Interventions: Other: Placebo
- Acute tryptophan depletion (Experimental): Amino acid drink without tryptophan. Ingested 4-5 hours prior to PET scanning.
  Interventions: Dietary Supplement: Acute tryptophan depletion

INTERVENTIONS:
Drug: Citalopram and Pindolol — Citalopram: selective serotonin reuptake inhibitor
  Pindolol: non-selective beta blocker and 5-HT1A receptor antagonist
  Other Names: Seropram; Hexapindol®
  Arms: Citalopram and Pindolol
Other: Placebo — On the second PET scanning day, subjects received a protein drink as well as a 50 ml saline infusion over 1 hour starting 30 min before PET scanning.
  Arms: Placebo
Dietary Supplement: Acute tryptophan depletion
  Other Names: Amino acid drink without tryptophan
  Arms: Acute tryptophan depletion

SUMMARY:
The purpose of this project was to introduce the recently developed positron emission tomography (PET) tracer [11C]Cimbi-36 for use in clinical studies and to investigate the ability of the tracer to quantify the 5-HT2A receptor in the human brain. As a receptor agonist, [11C]Cimbi-36 binding will provide a more functional picture of 5-HT2A receptors, while this binding is thought to be correlated to brain serotonin levels. Both measurement of signaling through the 5-HT2A receptor and measurement of serotonin levels in vivo would have great scientific relevance for significant diseases such as depression and schizophrenia.

DETAILED DESCRIPTION:
The serotonin 2A (5-HT2A) receptor is the most abundant excitatory serotonin (5-HT, 5-hydroxytryptamine) receptor in the human brain, and multiple positron emission tomography (PET) studies have investigated the 5-HT2A receptors in the human brain using antagonist radioligands. However, the currently available antagonist PET radioligands bind the total pool of 5-HT2A receptor receptors whereas a 5-HT2A receptor agonist binds the high-affinity subgroup of the receptors which are also G-protein coupled, and thus hypothesized to be the functional relevant population of receptors. At the Center for Integrated Molecular Brain Imaging (CIMBI), a novel agonist PET radioligands for brain imaging of 5-HT2A receptors was recently validated in animals (Ettrup et al. 2011, EJNMMI). In the human brain, [11C]Cimbi-36 was validated as a selective 5-HT2A receptor agonist PET radioligand through a blocking study with the 5-HT2A receptor antagonist pharmaceutical ketanserin. In this validation study, the biodistribution and kinetic modelling of [11C]Cimbi-36 binding in the human brain was also validated. With these studies, investigators will test the most promising of these, [11C]Cimbi-36, in clinical trials, where it will provide a novel method for detecting dysfunction in the 5-HT system. The specific aim of this clinical trial is:

- To examine the effect of acute alterations in 5-HT levels on cerebral [11C]Cimbi-36 binding in healthy volunteers who will be PET-scanned at baseline and after pharmacological or dietary interventions that either increase or decrease cerebral 5-HT levels.

It is hypothesized that this novel agonist radioligand will provide both a more physiological relevant measure of the 5-HT2A receptors and also reflect levels of cerebral 5-HT in humans, more specifically:

BP will decrease after pindolol and selective serotonin reuptake inhibitor (SSRI) treatment and increase after acute tryptophan depletion (ATD). Placebo will leave binding potential (BP) unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Generally healthy

Exclusion Criteria:

* primary psychiatric disorder
* current or previous neurological disease, severe somatic disease or taking medications that can influence the results.
* non-fluent in danish or severe visual or hearing impairment
* current or previous learning difficulties
* pregnancy or lactating
* contraindications for magnetic resonance scanning
* alcohol or drug abuse
* allergy to any of the used medications
* participation in studies with radioactivity (>10 mSv) within the last year or significant occupational exposure to radioactivity.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gitte M Knudsen, DMSc, Principal Investigator — Neurobiology Research Unit, Rigshospitalet
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Ettrup A, Hansen M, Santini MA, Paine J, Gillings N, Palner M, Lehel S, Herth MM, Madsen J, Kristensen J, Begtrup M, Knudsen GM. Radiosynthesis and in vivo evaluation of a series of substituted 11C-phenethylamines as 5-HT (2A) agonist PET tracers. Eur J Nucl Med Mol Imaging. 2011 Apr;38(4):681-93. doi: 10.1007/s00259-010-1686-8. Epub 2010 Dec 21. PMID 21174090

RESULTS

PARTICIPANT FLOW:
Groups:
- Citalopram and Pindolol: Citalopram intravenous infusion starting 30 min before scanning, 40 mg/h for 1 hour.
  Pindolol peroral administration starting 3 days before scanning:
  Day 1: 2.5 mg 3 times daily, day 2: 5 mg 3 times daily, day 3: 7.5 mg 3 times daily, Day 4 (scan day) 7.5 mg morning and noon.
  Citalopram and Pindolol: Citalopram: selective serotonin reuptake inhibitor
  Pindolol: non-selective beta blocker and 5-HT1A receptor antagonist
- Placebo: Placebo for pindolol: sugar tablets that resembles pindolol
  Placebo for ATD: amino acid drink balanced formula (containing tryptophan)
  Placebo for Seropram: NaCl infusion
  Placebo: On the second PET scanning day, subjects received a protein drink as well as a 50 ml saline infusion over 1 hour starting 30 min before PET scanning.
- Acute Tryptophan Depletion: Amino acid drink without tryptophan. Ingested 4-5 hours prior to PET scanning.
  Acute tryptophan depletion
Period: Overall Study
Arm/Group | Citalopram and Pindolol | Placebo | Acute Tryptophan Depletion
Started | 8 | 8 | 8
Completed | 8 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Citalopram and Pindolol | Placebo | Acute Tryptophan Depletion | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 24
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (2.1) | 22.6 (2.5) | 22.9 (3.2) | 22.6 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 4 | 4 | 4 | 12
Region of Enrollment [Number; unit: participants]
  Denmark | 8 | 8 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Neocortical [11C]Cimbi-36 BPND From Baseline to Intervention in Each Arm
Description: Cerebral Cimbi-36 receptor binding is measured with PET scanning for 2 hours, at baseline and after intervention. The resultant time-activity curves for brain tissue are used together with time-activity curves obtained with blood samples and kinetic modelling to yield unitless values of BPND at baseline and after intervention, respectively. As outcome, the mean percent difference from baseline to intervention in each arm is measured.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Citalopram and Pindolol | Placebo | Acute Tryptophan Depletion
Number analyzed (Participants) | 8 | 8 | 7
percent change | 7.4 (16) | 0.6 (7.2) | 3.8 (0.2)

ADVERSE EVENTS:
Arm/Group | Citalopram and Pindolol | Placebo | Acute Tryptophan Depletion
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram and Pindolol (N=8) | Placebo (N=8) | Acute Tryptophan Depletion (N=8)
AE (General disorders) | 0 (0) | 0 (0) | 1 (1) — Anaphylactic reaction

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No